CLINICAL TRIAL: NCT05012566
Title: Clinical, Instrumental and Histological Evaluation of the Combined Use of Onabotulinumtoxin A and Hyaluronic Acid Fillers in Patients With Facial Paralysis
Brief Title: Onabotulinumtoxin A and Hyaluronic Acid Fillers in the Treatment of Facial Paralysis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Dario Bertossi, Prof., Department of Chirurgia Maxillo-Facciale and Odontostomatologia, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FACIAL PARALYSIS
Record Dates: First submitted 2021-06-25; First posted 2021-08-19 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Hemifacial Paralysis
MeSH Terms: conditions — Facial Paralysis | interventions — Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Intervention Model Description: monocenter, no treated controlled group, randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyaluronic Acid filler and Botulinum Toxin group (Experimental): 1. Hyaluronic Acid filler:
     * Juvederm Volbella: it will be used in the softer soft tissue, beacuse its reology is the softest
     * Juvederm Volift: it will be used in malar area, because its reology is intermediate between the three products
     * Juvederm Voluma: il will be used unstructured area bacause it has the best rheologic characteristics in the reintegration of loss of tissue.
     The differents products are going to use in different areas, depending on the area of the paralysis.
  2. Botulinum Toxin:
     * Vistabex (50U/vial): it is going to be used in the controlateral area of the paralysed face, in order to relax muscle hyper-tonicity.
  Dosage and administration steps will be selected according to the clinical situation.
  Interventions: Device: Juvederm; Drug: Vistabex
- Control group (No Intervention): The control group will undergo at the same examinations of the treated group but it will not be subjected to any treatment.

INTERVENTIONS:
Device: Juvederm — * Juvederm Volbella: 15mg/ml, it is injected 1.5ml per patient per treatment (a total of 3ml per patient split in 2 treatment sessions at a 4 months interval);
  * Juvederm Volifit: 17.5mg/ml, it is injected 3ml per patient per treatment (a total of 6ml per patient split in 2 treatment sessions at a 4 months interval);
  * Juvederm Voluma: 20mg/ml, it is injected 5ml per patient per treatment (a total of 10ml per patient split in 2 treatment sessions at a 4 months interval)
  Other Names: Hyaluronic Acid
  Arms: Hyaluronic Acid filler and Botulinum Toxin group
Drug: Vistabex — Vistabex: 50U/vial, it is injected up to 80U per patient per treatment (2 treatment sessions at a 4 months interval)
  Other Names: Botulinum Toxin
  Arms: Hyaluronic Acid filler and Botulinum Toxin group

SUMMARY:
Social interaction via facial mimic expression is crucial in human relationship and communication. Neural function disorder in this mechanism therefore affects human communication and social interaction. Facial nerve palsy is the paralysis of any structure innervated by the facial nerve, thus inibiting and severely compromising facial expression. In the last decade a new algorithm of treatment of facial paralysis has been raised. It connects the expertise of Aesthetic Medicine with the expertise of Plastic and Reconstructive Surgery. It is based on the use of Botulinum Toxin (BT) and Hyaluronic Acid (HA fillers). Botulinum toxin is a paralytic toxin that determine flaccid paralysis and is nowadays used in the static correction of facial paralysis with minimal invasiveness, optimal results and no time consumption. The HA fillers has the ability to restore facial volume loss and it is used in the treatment of facial palsy to harmonize symmetry. The aim is to study the effects of the BT and HA in facial paralysis patients in order to understand the efficacy of these products that have never been injected together in this type of patients. Primary objective. To evaluate the functional improvement of facial asymmetries due to facial nerve lesion after the treatment with OnabotulinumtoxinA and hyaluronic acid fillers compared with the untreated group. The evaluation will be performed analyzing the two groups at the baseline (visit 0) and the end of the treatment period (visit 5, after 9 months). Improvement difference of at least 1 grade on the House-Brackmann scale, compared with the untreated group, will be considered clinically significant. Methods. The investigation is randomized open lab phase II single centre clinical trial. This experimental study proposes to evaluate a group of 70 patients affected by hemifacial paralysis of level 3 to 6 on the House-Brackmann scale. 35 patients will be treated (Group A) with both OnabotulinumtoxinA and hyaluronic acid fillers with a monitored follow up. A control group of 35 patients (Group B) who will not be treated, will be enrolled to compare the efficacy of the treatment. During the study all the AE/ADR will be recorded.

DETAILED DESCRIPTION:
The patients will be evaluated with instrumental (3D pictures, neuro-physiological examination (EMG), radiological [Magnetic Resonance Imaging (MRI)], Cone Beam Computer Tomography (CBCT) and Ultrasound (US)) and non-instrumental analysis (clinical questionnaires and hystological analysis). The histology will be performed with both traditional and electronic approaches. The area of the biopsy will be the paralytic area in the two groups in order to study the soft tissue modulation of the injected molecules. Patient's qiality of life (QoL), through specifically test (FACE-Q), will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > 18 years and < 65 years
2. Hemifacial paralysis from 3 to 6 on the House-Brackmann scale
3. Never treated with HA and BTX injection
4. Signed informed consent
5. Women of childbearing potential will only be included in the study if uptaking hightly effective birth control measures.

Exclusion Criteria:

1. Hypersensitivity to any component of the products used
2. Diabetes, systemic disease, coronary artery disease, acute-chronic hepatitis C, autoimmune disease and/or other disease involving poor general health clotting problem. Peripheric neuro-musculars disorders, amyotrophic lateral sclerosis.
3. Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2023-07-14 (Estimated); Study Completion 2023-07-14 (Estimated)

PRIMARY OUTCOMES:
House-Brackmann scale | Day 0 and day 270
  Change from baseline House-Brackmann score at day 270 will be assessed and then compared between the trial groups. The House-Brackmann score is a score to grade the degree of nerve damage in a facial nerve palsy.
  The measurement is determined by measuring the upwards (superior) movement of the mid-portion of the top of the eyebrow, and the outwards (lateral) movement of the angle of the mouth. Ti is consist of VI level: Grade I - Normal; Grade II - Slight Dysfunction; Grade III - Moderate Dysfunction; Grade IV - Moderate Severe Dysfunction; Grade V - Severe Dysfunction; Grade VI - Total Paralysis

SECONDARY OUTCOMES:
Facial Appearance | Day 0 and day 270.
  Facial Appearance will be assessed by FACE-Q Appearance scale measuring different concepts: Area Under Chin, Cheeks, Crows' Feet, Eyes, Forehead & Eyebrows,Lines Between Eyebrows, Lip Lines, Lower Eyelids, Marionette Line, Neck, Nostrils, Upper Eyelids, Cheekbones, Chin, Eyelashes, Face Overall, Forehead Lines, Lines Overall, Lips, Lower Face & Jawline, Nasolabial Folds, Nose, Skin.
  Each scale is composed of a series of items (or questions) that evaluate a concept of interest. Patient responses to items are on a four-point scale and are asked to answer with their face/facial appearance in mind. Answers for a scale are summed and converted to a score from 0 to 100. A higher score indicates a better outcome.
Health-Related Quality of Life | Day 0 and day 270
  Health-Related Quality of Life will be assessed by FACE-Q Quality of Life scale measuring different concepts: Age Visual Analogue (score ranging from -15 to +15), Aging Appraisal, Appearance-Related Distress, Early Life Impact of Treatment, Expectations, Psychological Function, Recovery Early Symptoms, Decision Satisfaction, Outcome Satisfaction,Social Function.
  Each scale is composed of a series of items (or questions) that evaluate a concept of interest. Patient responses to items are on a four-point scale. Answers for a scale are summed and converted to a score from 0 to 100. For most of these scales, a higher score indicates a better outcome.
Adverse Effects | Day 0 and day 270
  Adverse Effects related to different parts of the face (Cheeks, Lower Face, Neck, Eyes, Forehead, Eyebrows, Scalp, Lips, Nose, Skin) will be assessed by FACE-Q Adverse Effects scales.
  Each scale is composed of a series of items (or questions) that evaluate a parts of the face. Patient responses to items are on a three/four-point scale. Answers for a scale are summed and converted to a score from 0 to 100. A higher score indicates a better outcome.
Patients experience of care | Day 0 and day 270
  Patients experience of care related to satisfaction with information, medical team, office staff and with doctor/surgeon will be assessed by FACE-Q experience of care scales.
  Each scale is composed of a series of items (or questions) that evaluate the satisfaction. Patient responses to items are on a four-point scale. Answers for a scale are summed and converted to a score from 0 to 100. For all these scales, a higher score indicates a better outcome.
Facial symmetry | Day 0, day 20, day 150, day 270
  Facial symmetry will be performed through the analisys of 3D-photography implemented with a face grid, that allows the quantification of symmetry of the face. The face grid permits to calculate the distance in millimeters of two points from the midline (both in vertical and horizontal direction).
Facial aesthetic | Day 0 and day 270
  Facial aesthetic will be evaluated through the analysis of 3D-photography implemented with a face grid and the Arnett's aesthetic analysis, in order to appreciate the improvement of facial aesthetic.
Facial aesthetic - thickness of soft tissue | Day 0 and day 270
  The thickness of soft tissue will be evaluated using MRI and US (millimetric quantification of the thickness of different areas)
Facial aesthetic - thickness of hard tissue | Day 0 and day 270
  The thickness of hard tissue will be evaluated using CBCT (millimetric quantification of the thickness of the different areas)
Facial aesthetic - tropism of muscles | Day 0 and day 270
  The tropism of muscles will be evaluated using US and cathegorized in atrophy, hypotrophy, eutrophy, hypertrophy.
Facial aesthetic - patho-physiological condition | Day 0 and day 270
  The patho-physiological condition will be evaluated throught an histological analysis that provides a qualitative analysis of injected and not injected tissue and specifically the effects on the fiber muscles
Hystological analysis | Day 0 and day 270
  % of patients with tissue changes assessed by hystological analysis using scanning electron microscope and/or transmission electron microscope provides a through examination of tissue changes due to the physical introduction of the products, comparing different conditions in injected and not-injected tissue and eventually any effect on the fiber muscles.
EMG | Day 0 and day 270
  EMG provides eletric potentials of the facial neuromuscular complex in order to evaluate the activity and symmetry oh their function.
Adverse Events | Day 0, day 20, day 30, day 140, day 150, day 270
  Registration of number and type of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dario Bertossi, Prof, Principal Investigator — AOUI Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata, Verona, Italy

IPD SHARING:
Plan to Share IPD: No